CLINICAL TRIAL: NCT05116462
Title: A Randomized, Double-blind, Phase 3 Study of the Efficacy and Safety of Sindilizumab Combined With Chemotherapy or Placebo Combined With Chemotherapy for Neoadjuvant and Adjuvant Therapy for Resectable Non-small Cell Lung Cancer (ORIENT-99)
Brief Title: Neoadjuvant and Adjuvant Therapy Studies of Sindilizumab in Resectable Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI308G301
Record Dates: First submitted 2021-10-26; First posted 2021-11-11 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Paclitaxel; sintilimab; Cisplatin; Taxes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sintilimab (Experimental): Neoadjuvant Treatment period: up to 3 cycles of sintilimab plus platinum-based chemotherapy prior to surgery.
  adjuvant Treatment period: Subjects will receive 1 cycle of sintilimab plus platinum-based chemotherapy, and then receive sintilimab therapy after surgery until disease recurrence, unacceptable toxicity, receiving new anti-tumor therapy, withdrawal of informed consent (ICF), lost to follow-up or death, or other conditions that require treatment discontinuation (whichever occurs first). The maximum duration of postoperative treatment with either sintilimab or placebo is 13 cycles.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Sintilimab; Drug: Cisplatin; Drug: Nab paclitaxel
- Placebo (Placebo Comparator): Neoadjuvant Treatment period: up to 3 cycles of placebo plus platinum-based chemotherapy prior to surgery.
  adjuvant Treatment period: Subjects will receive 1 cycle of placebo plus platinum-based chemotherapy, and then receive placebo therapy after surgery until disease recurrence, unacceptable toxicity, receiving new anti-tumor therapy, withdrawal of informed consent (ICF), lost to follow-up or death, or other conditions that require treatment discontinuation (whichever occurs first). The maximum duration of postoperative treatment with either sintilimab or placebo is 13 cycles.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin; Drug: Nab paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 D1 IV Q3W
Drug: Carboplatin — AUC 5 or 6 mg/ml/min D1 IV Q3W
Drug: Paclitaxel — 175 or 200 mg/m2 D1 IV Q3W
Drug: Sintilimab — 200 mg D1 IV Q3W
  Arms: Sintilimab
Drug: Cisplatin — 75 mg/m2 D1 IV Q3W
Drug: Nab paclitaxel — 100 mg/m2 D1, 8, 15 IV Q3W
Drug: Placebo — 20 ml D1 IV Q3W
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind Phase 3 study to compare the efficacy and safety of Sindilizumab combined with chemotherapy or placebo combined with chemotherapy for neoadjuvant and adjuvant therapy for Resectable Stage II to IIIB (resectable N2 only) non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign the written informed consent form (ICF), and be able to follow the visits and relevant procedures specified in the protocol.
2. Age ≥ 18 years.
3. Cytologically or histologically confirmed primary NSCLC (including adenocarcinoma, squamous cell carcinoma).
4. Subjects with Stage II, IIIA or IIIB (resectable N2 only) disease based on the 8th edition of the TNM staging classification for lung cancer issued by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification (AJCC8).
5. Deemed radically resectable with curative intent.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
7. Have not received any prior systemic anti-tumor therapy or local radiotherapy for NSCLC.

Exclusion Criteria:

1. Subjects with confirmed or suspected brain metastases.
2. Currently participating in an interventional clinical study or treatment with another study drug or study device within 4 weeks prior to randomization.
3. Received Chinese herbal medicine, Chinese traditional medicine with anti-tumor indications, or drugs with immunomodulatory effects (including thymosin, interferon, interleukin) within two weeks prior to randomization
4. Received a live attenuated vaccine 4 weeks prior to randomization (or planned to receive a live attenuated vaccine during the study).
5. Requiring long term systemic corticosteroids
6. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive), known active syphilis.
7. Active hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-10-14 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) in stage III NSCLC | Up to approximately 2 years following the beginning of Post-operative Assessment baseline(up to Study 2 years )
  Up to approximately 2 years following the beginning of Post-operative Assessment baseline(up to Study 2 years )
Event Free Survival (EFS) in ITT population | Up to approximately 3 years following the beginning of Post-operative Assessment baseline(up to Study 3 years )
  EFS is defined as the time from randomization to the first recorded time to any first documented progression, recurrence or death, which occurs first.

SECONDARY OUTCOMES:
Disease free survival (DFS) | Up to approximately 2 years following the begining of Post-operative Assessment baseline(up to Study 5.4 years )
  DFS is defined as the time from surgery to disease recurrence or death due to any cause.
Major Pathological Response (mPR) Rat | Up to approximately 6 weeks following completion of neoadjuvant treatment (up to Study 2 years)
  mPR rate is defined as ≤ 10% residual invasive viable tumor in both the primary tumor (lung) and the sampled lymph nodes after neoadjuvant therapy.
Overall survival (OS) | Up to approximately 5.4 years
  OS is defined as the time from randomization to death due to any cause.
Safety parameters:AE | Up to approximately 5.4 years
  The relationship of study drug and the severity of all adverse events (AEs), treatment emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), immune-related adverse events (irAEs), serious adverse events (SAEs), infusion-related reactions (IRRs) and surgery delay rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China